CLINICAL TRIAL: NCT05964673
Title: Effect of Bioptron Light Therapy on Dryness of Eyes in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004549
Record Dates: First submitted 2023-07-18; First posted 2023-07-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Postmenopausal Women

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- education program group (No Intervention): this group will receive patient education program for four weeks.
  1. limiting screen time
  2. blinking awareness training
  3. keeping the home environment cool and moist
  4. using artificial tears (Hylo®gel) twice daily
  5. contact lens use can preferably be limited,
  6. adding omega-3 poly unsaturated fatty acids in the diet or as dietary supplements.
- bioptron light therapy group (Experimental): Patients will be sitting in a comfortable chair, with their eyes closed, with cleaned eyelids, and occasionally blinking. Bioptron lamp will be lined at an angle of 90°, at a distance from 5 cm to 10 cm, exposure time will be 5 min. Energy is very low, 1 - 2.4 J/cm without thermal effects, energy density is 40mW. Bioptron light is polychrome, wave frequency is from 400 nm (including blue, visible radiation) up to 2000 nm (representing infrared waves)
  Interventions: Device: bioptron light therapy

INTERVENTIONS:
Device: bioptron light therapy — patients will receive patient education program and bioptron light therapy for four weeks
  Arms: bioptron light therapy group

SUMMARY:
Dry eye disease (DED) is a growing public health concern affecting quality of life and visual function, with a significant socio-economic impact. It is more prevalent in the females and is being specifically in the menopausal and postmenopausal age group.

Bioptron light therapy is efficient in the elimination of allergic reactions, signs and symptoms of dry eye improving capillary circulation, immunity stimulation, relieving pain and establishing balance of tissue electromagnetic field

DETAILED DESCRIPTION:
Around 60 postmenopausal women will be randomly divided into two equal groups, they all complain from dry eye symptoms, ranging from mild/normal to moderate and severe.

Group(A): will receive patient education program for four weeks. Group(B): will receive patient education program and bioptron light therapy for four weeks

ELIGIBILITY:
Inclusion Criteria:

* All participants are postmenopausal women.
* Their age above 50 years old
* All participants aren't on any systematic therapy.

Exclusion Criteria:

* • Injuries and previous surgical treatment of eyes

  * All patients with diagnosis of chronic blepharitis, meibominitis or any other eye infections
  * Participants with autoimmune diseases such as Sjögren's syndrome (SS), rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE)
  * Diabetic participants will be excluded.
  * Smokers will be excluded from the study.
  * The use of Hormone Replacement Therapy

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-09-19 (Estimated); Study Completion 2023-11-08 (Estimated)

PRIMARY OUTCOMES:
Dry Eye-Related Quality-Of-Life Score (DEQS) | Dry Eye-Related Quality-Of-Life Score will be measured at baseline, and it will be measured again after four weeks
  The Dry Eye-Related Quality-Of-Life Score questionnaire is a 15-item instrument for assessing subjective dry eye symptoms and their effects on activities of daily living within the previous week.
  1. extremely good
  2. very good
  3. good
  4. bad
  5. very bad
  6. extremely bad
Tear Breakup Time (TBUT) | Tear Breakup Time will be measured at baseline, and it will be measured again after four weeks
  Tear Breakup Time Is the time interval between a complete blink and the appearance of the first break, discontinuity or dry spot observed in the tear film.

SECONDARY OUTCOMES:
Schirmer's test | Schirmer's test will be measured at baseline, and after four weeks
  The Schirmer test score is determined by the length of the moistened area of the strips (using the scale packaged with the strips) and the duration of the measurement in minutes. A score of greater than 10 mm in 5 minutes is accepted as normal. A score of less than 5 mm in 5 minutes indicates a tear deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ahmed, lecturer, Principal Investigator — giza, Egypt, 12511
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Mohamed Elsayed Saad E, Magdy Ahmed S, Mohamed Yousef A, Shahat Hassan E. Effect of Bioptron light therapy on dryness of eyes in postmenopausal women: a randomized controlled trial. Lasers Med Sci. 2026 Feb 4;41(1):20. doi: 10.1007/s10103-026-04807-6. PMID 41634440